CLINICAL TRIAL: NCT03652649
Title: Evaluation of Efficacy and Safety of Ketogenic Complete Meal Replacement as Treatment of Obesity-related Type 2 Diabetes Mellitus
Brief Title: Treatment of Type 2 Diabetes With Ketogenic Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mid-Atlantic Epilepsy and Sleep Center, LLC (Other)
Responsible Party: Principal Investigator, Pavel Klein, Principal Investigator, Mid-Atlantic Epilepsy and Sleep Center, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: maes 009
Record Dates: First submitted 2018-07-05; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Type2 Diabetes Mellitus; Obesity
Keywords: type 2 diabetes; diabetes; ketogenic diet; low carb diet; weight loss; obesity; diet treatment; nutrition; BMI
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3:1 Ketogenic Complete Meal Replacement (Experimental): Evaluating glycemic control and weight loss in obese participants with type 2 diabetes treated for 6 months with 3:1 [fat]:[protein+carbohydrate] ratio, 1600 kcal/day complete meal replacement ketogenic diet
  Interventions: Other: 3:1 ratio Ketogenic diet

INTERVENTIONS:
Other: 3:1 ratio Ketogenic diet — Type 2 Diabetic subjects with BMI greater than or equal to 30 are started on 3:1 ratio ketogenic complete meal replacement program and weight loss and glycemic control is tracked over 6 month intervention period
  Other Names: Classic Ketogenic Diet

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of ketogenic diet (KD) complete meal replacement treatment of obesity-related Type 2 diabetes mellitus (T2DM) and of obesity in patients with obesity and T2DM. This will be an open-label single arm study evaluating glycemic control and weight loss in obese participants with type 2 diabetes treated for 6 months with 3:1 [fat]:[protein+carbohydrate] ratio, 1600 kcal/day diet.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy and safety of ketogenic diet (KD) complete meal replacement treatment of obesity-related Type 2 diabetes mellitus (T2DM) and of obesity in patients with obesity and T2DM. This will be an open-label single arm study evaluating glycemic control and weight loss in obese participants with type 2 diabetes treated for 6 months with 3:1 [fat]:[protein+carbohydrate] ratio, 1600 kcal/day diet.

Treatment will consist of KD complete meal replacement with 3:1 [fat]: [protein + carbohydrate] weight ratio, and with 1600 kcal restriction. It will consist of pre-made meals, including breakfast, lunch, dinner and two snacks, one each between breakfast and lunch and lunch and dinner. Meals will be made according to supplied recipes (Anemone, LLC.) with a 3-week long meal plan consisting of different recipes for the 3 meals and 2 snacks different for each day of the 3-week cycle, with repeating cycles. All KD-treated participants will receive the same meal plan. Meals will be prepared uniformly by one facility and will be delivered to participants frozen once a week in packages subdivided into individual days with each day's package containing 5 separately packaged meals. Participants will be given a list of allowed 0 calories drinks and will consume no non-allowed beverages. Reductions to oral glycemic medications will occur at the start of the diet.

Participants will be evaluated in face-to-face visit during weeks 1, 2 and 4 of the study, then monthly (see Table 1, visit schedule). Evaluations will include weight, BMI, BP, waist circumference, adverse events and treatment compliance. Participants will check their blood glucose levels 3x/day, including am fasting, mid-day and evening 2 hours post-prandial, and urine for ketones levels with Ketostix (Bayer AG, IN, U.S.A.) 2x/day. They will record results in a glucose and ketone level diary which will be reviewed at each visit. Laboratory evaluations will include 8 am serum fasting glucose, insulin levels, C-peptide and lipid panel, HbA1C, serum beta-hydroxybutyrate (BOH), leptin levels, C-reactive protein (CRP), complete blood count (CBC), basic metabolic profile (BMP), renal and liver functions tests (LFTs), and uric acid. Laboratory evaluations will be obtained once at baseline prior to treatment initiation, at 3 and 6 months after treatment initiation. Hunger will be evaluated with a 7-point Likert scale (range: extremely hungry to extremely full) which will be administered at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70
2. Ability and willingness to sign informed consent form.
3. T2D with BMI ≥ 30 kg/m2
4. Stable hypoglycemic medications for at least 2 months

Exclusion Criteria:

1. History of bariatric surgery ≤ 2 years prior to enrollment.
2. Any systemic illness or unstable medical condition that might pose additional risk, including: cardiac, unstable metabolic or endocrine disturbances, renal or liver disease, past history of renal calculi, hyperuricemia, hypercalcemia, mitochondrial disease, known disorder of fatty acid metabolism, porphyria, and active systemic cancer.
3. History of uncontrolled hyperlipidemia
4. Change in the dose or type of hypoglycemic treatment within 1 month prior to enrollment.
5. Psychosis within six months of enrollment, evidenced by treatment with anti-psychotic medications with recent medication initiation or dose increase.
6. Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators would interfere with adherence to study requirements;
7. History of cerebrovascular disease or unstable heart disease within 6 months of enrollment
8. Pregnancy
9. Use of any investigational drugs within 3 months of enrollment.
10. Inability or unwillingness of subject to give written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Type 2 diabetes remission | 6 months (study duration)
  Defined as normal fasting blood glucose (<126), normal HbA1C (<6.4%), and no diabetic medications

SECONDARY OUTCOMES:
Change from baseline in glucose blood level in patients with type 2 DM in 6 months. | 6 months (study duration)
  Defined as normal fasting blood glucose (<126), normal HbA1C (<6.4%), and no diabetic medications
Percentage of diabetic medication load reduction | 6 months (study duration)
  Change in diabetic medication load
Change from baseline in HbA1C in patients with type 2 DM in 6 months. | 0, 3 and 6 months treatment duration
  HbA1C
Adverse events | 6 months (study duration)
  Adverse events occurrence
Fasting serum insulin | 0, 3 and 6 months treatment duration
  Change in fasting serum insulin value
BMI | Day 0, Day 7, Day 14, Month 1, 2, 3, 4, 5 and 6
  Change BMI from baseline
Weight | Day 0, Day 7, Day 14, Month 1, 2, 3, 4, 5 and 6
  Change weight from baseline
Waist circumference | Day 7, Day 14, Month 1, 2, 3, 4, 5 and 6
  Change waist circumference from baseline
Blood pressure | Day 7, Day 14, Month 1, 2, 3, 4, 5 and 6
  Change of systolic and diastolic blood pressures from baseline
Urine ketone levels | Day 7, Day 14, Month 1, 2, 3, 4, 5 and 6
  Urine ketone levels evaluation
Fasting leptin levels | 0, 3 and 6 months treatment duration
  Fasting leptin levels evaluation
Fasting lipid levels | 0, 3 and 6 months treatment duration
  Fasting lipid levels evaluation
Hunger scale scores | Day 0, Day 7, Day 14, Month 1, 2, 3, 4, 5 and 6
  Likert scale (range: extremely hungry to extremely full) which will be administered at each visit.The best outcome is 5=satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Klein, M.B,B.Chir., Principal Investigator — Mid-Atlantic Epilepsy and Sleep Center
Locations (1):
- Ivana Tyrlikova, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No